CLINICAL TRIAL: NCT03855748
Title: Hip Peak Torque in Running and Jumping Activities in Healthy Active Subjects - a Cross-Sectional Study
Brief Title: Hip Peak Torque in Running and Jumping Activities in Healthy Active Subjects
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Ishøi, Principal Investigator, Hvidovre University Hospital
Other Study IDs: Hip Biomechanics
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Healthy group — Subjects undergo the following activities:
  1. Walking
  2. Jogging (8-11 km/h)
  3. Maximal 5 meters sprint acceleration
  4. Single leg drop jump from 35 cm height
  5. Horizontal jump with single leg landing with a distance of 100% and 150% of leg length
  6. Maximal change of direction at 45, 135, 180 degrees
  7. Single-leg cross-country skiing exercise

SUMMARY:
Hip-related groin pain is common in sports that involves change of direction, kicks and sprint accelerations such as football, ishockey, tennis and basketball. Groin pain symptoms either pre- or post-treatment may be load-related, there is limited information on how different sporting activities affect hip joint loading. Thus, the purpose of this explorative cross-sectional study is to investigate hip peak torque in running and jumping activities in healthy active subjects.

Such information may guide furture rehabilitation strategies and return to sport sport criteria.

Twenty healthy subjects from the Capital Region of Denmark with an age of 18-40 will be included.

Hip joint kinetics and kinamatics will be obtained during the following activities for each subjects:

1. Walking
2. Jogging (8-11 km/h)
3. Maximal 6 meters sprint acceleration
4. Single leg drop jump from 35 cm height
5. Horizontal jump with single leg landing with a distance of 100% and 150% of leg length
6. Maximal change of direction at 45, 135, 180 degrees
7. Single-leg cross-country skiing exercise

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are healthy and physically active.

Exclusion Criteria:

* Any history of lower limb surgery or fracture
* Lower limb injuries, joint or muscle pain with a duration of more than 6 weeks within the past year.
* Body Mass Index more than 30 kg/m2

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-03-24 (Actual)

PRIMARY OUTCOMES:
Hip peak torque, Nm/kg | Baseline (week 0)
  Hip peak torque (Nm/kg) measured in the following activities:
  1. Walking
  2. Jogging (8-11 km/h)
  3. Maximal 5 meters sprint acceleration
  4. Single leg drop jump from 35 cm height
  5. Horizontal jump with single leg landing with a distance of 100% and 150% of leg length
  6. Maximal change of direction at 45, 135, 180 degrees
  7. Single-leg cross-country skiing exercise

SECONDARY OUTCOMES:
Angle at peak torque, degrees | Baseline (week 0)
  Angle at hip peak torque (degrees) measured in the following activities:
  1. Walking
  2. Jogging (8-11 km/h)
  3. Maximal 5 meters sprint acceleration
  4. Single leg drop jump from 35 cm height
  5. Horizontal jump with single leg landing with a distance of 100% and 150% of leg length
  6. Maximal change of direction at 45, 135, 180 degrees
  7. Single-leg cross-country skiing exercise

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Ishøi, PhD student, Principal Investigator — Sports Orthopedic Research Center - Copenhagen (SORC-C)
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided